CLINICAL TRIAL: NCT03743623
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Neurocytotron in Patients With Cerebral Palsy
Brief Title: Neurocytotron on Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurocytonix, Inc. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCX-CP-01
Record Dates: First submitted 2018-11-09; First posted 2018-11-16 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Study treatment with Neurocytotron, which is a device is designed to generate a controlled beam of electromagnetic waves of certain frequencies in the presence of a magnetic field with pre-determined strength.
  Interventions: Device: Neurocytotron
- Placebo Group (Placebo Comparator): The placebo control is a mock treatment in which a subject will go through the same procedures as subjects assigned to the treatment group, only without being actually exposed to electromagnetic waves and magnetic fields.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Neurocytotron — Neurocytotron utilizes a combination of instantaneous magnetic field and low-spectrum radiofrequency waves for therapeutic purpose. Its working principle is based on the theory of magnetic resonance.
  Arms: Treatment Group
Device: Placebo — Same treatment procedures without being actually exposed to electromagnetic waves and magnetic field
  Arms: Placebo Group

SUMMARY:
This is a randomized, double-blinded, two-arm, placebo-controlled clinical study. The enrollment will be randomized 1:1 to Neurocytotron treatment or mock treatment (placebo).

Upon the completion of the study period, the placebo group will receive treatment, if the study results show benefits to patients.

DETAILED DESCRIPTION:
The study proposes to investigate the use of non-thermal and non-radioactive radiofrequency pulses in the brain for improving the symptoms of cerebral palsy. The proposed treatment will deliver radiofrequency pulses to the brain of patients in a non-invasive manner. The duration of the treatment will be 1 hour per day, for 28 days. After treatment, participants will be monitored for two months to detect potential adverse events and any signs of symptoms improvement. The study will be closed once 48 subjects complete the study. At the end of the study, the placebo group will have the opportunity to receive treatment with the Neurocytotron, based on the benefits shown by study results.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Form approved by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) signed and dated by the subject or the subject's legal representative and by the Principal Investigator. This must be obtained before the performance of any study-related procedures that are not part of normal participant care.
2. Patients 1 to 8 years old (We will include this age range because children with CP less than 1-year-old have a high mortality rate, in addition, the clinical evolution stabilizes after the second year of life, and the potential effect of treatment is optimized in the first 5 years).
3. A clinical diagnosis of spastic cerebral palsy, or spastic and dyskinetic, secondary only to hypoxic/ischemic encephalopathy
4. For spasticity, having scored at least 3 on the Ashworth scale, and 3 on the gross motor scale.
5. For dyskinesis, any degree.

Exclusion Criteria:

1. Patient with diagnosis of ataxia.
2. Current or recent history (within 2 months) of significant bacterial, fungal, viral, or mycobacterial infection.
3. Having a condition considered as causing or likely to cause co-morbidities, as determined by the investigator based on medical history, physical examination, vital signs, and clinical laboratory tests.
4. Subject with magnetic implants, pacemakers, claustrophobia or any other condition that precludes them from entering or staying in the NeuroCytotron.
5. Surgical history related to spasticity treatment.
6. Patients who have received treatment with botulinum toxin in the last 6 months.
7. 7. Children with prior neurosurgery within the past 6 months at the time of evaluation.
8. History of malignancy.
9. History of congenital heart disease.
10. Subjects who cannot or are unlikely able to comply with the protocol, according to the consensus reached by the group of study investigators.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | 28 Days
  Using Pediatric Evaluation of Disability Intervention (PEDI) and Pediatric Quality of Life Inventory (PedsQL) Scales
Spasticity | 28 Days
  Using Ashworth Scale from Baseline and Gross Motor Scale from Baseline

SECONDARY OUTCOMES:
Reduction in Use of Baseline Drug Treatment | 28 Days
  Compared to Placebo Group
Decreases in Use of Orthoses | 28 Days
  Compared to Placebo Group
Reductions in Number of Seizures or Epileptic Crisis | 28 Days
  Compared to Placebo Group
Changes in functional activity and brain anatomy | 28 Days
  Using functional Magnatic Resonance Imaging (fMRI), Diffusion Tensor Imaging (DTI) and Electroencephalography (EEG)
Evaluation of Adverse Events | 28 Days
  Compared to Placebo Group

CONTACTS AND LOCATIONS:
Overall Officials: J. Roberto Trujillo, MD, ScD, Study Chair — Neurocytonix, Inc.; Lorenzo R Morales Mancías, MD, Principal Investigator — NeuroCytonix México
Locations (1):
- NeuroCytonix México, Monterrey, San Pedro Garza García, Mexico

IPD SHARING:
Plan to Share IPD: No